CLINICAL TRIAL: NCT00773708
Title: Pilot Study to Assess the Role of Immune Activation and Apoptosis as a Marker for Treatment Intensification With Raltegravir in Hiv-infected Patients on Antiretroviral Therapy With Long-term Viral Suppression and Unfavourable Immunologic Response (Discordant Patients: v+i-)
Brief Title: Pilot Opened Trial in HIV-infected Patients Including an Investigational Marketed Product
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Sílvia Gel, Eugenia Negredo, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DISCOR-RAL
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2011-09

CONDITIONS: HIV Infections
Keywords: HIV infection; Discordant patient; CD4 recovery; intensification antiretroviral therapy; raltegravir; HIV-1 infected patient classified as "discordant" who showed high level of CD8+HLADR+CD38+ and cell death values at the screening
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): intensify their triple-drug therapy with Raltegravir (RAL)
  Interventions: Drug: raltegravir
- 2 (No Intervention): Continue with the same antiretroviral therapy

INTERVENTIONS:
Drug: raltegravir — intensify their therapy with Raltegravir(RAL):1 Protease inhibitor plus 2 nucleoside reverse transcriptase inhibitor plus RAL or 1 non-nucleoside reverse transcriptase inhibitor plus 2 nucleoside reverse transcriptase inhibitor plus RAL
  Other Names: N/P.
  Arms: 1

SUMMARY:
This study aims to provide new knowledge about the pathogenesis of HIV infection, specifically, the role that immune activation and apoptotic activity play in immune recovery, and in particular, in the paradoxical immunologic response of some patients on antiretroviral therapy despite achievement of sustained and complete viral suppression. In this regard, the investigators will prospectively evaluate the impact of intensification with Raltegravir in those "discordants" patients with high index of immune activation, measured as the percentage of CD8+HLADR+CD38+ cells. This will provide relevant information on the effectiveness of this drug in guided intensification regimens.

DETAILED DESCRIPTION:
One of the many adverse consequences of the human immunodeficiency virus (HIV) infection is the increase in the rate of lymphocyte cell death (Badley AD, Blood. 2000; 96:2951-64). Increased lymphocyte death is associated with the level of activation of the immune system (Gougeon ML. Nat Rev Immunol. 2003: 3:392-404), along with the disregulation of the cytokine network and a plethora of cytotoxic effects induced by HIV proteins (Badley AD, Blood. 2000; 96:2951-64). Hence, cell death can be observed in vivo not only in CD4+ cells, which are the main target of HIV, but also in CD8 T cells. Current knowledge suggest that immune activation and different mechanisms of cell death play a determinant role in T-lymphocyte (CD4+) loss during HIV infection and recovery after HAART (Bofill M et al AIDS. 1996 :827-34).

Highly active antiretroviral treatment (HAART) induces a decline in the level of immune activation and lymphocyte apoptosis in HIV-infected patients as a result of a reduction in viral replication (Kolber MA, et al, Clin Immunol. 2007 [Epub ahead of print]). This reduction contributes to the recovery of immune system associated with antiretroviral therapy. In addition to this effect, which is induced through the reduction in viral load, antiretroviral therapy has been implicated in the regulation of apoptosis in different cell types, inhibiting or activating the process and influencing treatment efficacy and toxicity (Petit F, et al.Trends Pharmacol Sci. 2005. 26:258-64).

Interestingly, it is not always true that antiretroviral therapy and viral suppression are associated with progressive immune recovery. Approximately 30% of patients present a paradoxical response to treatment, achieving progressive increases in immunity (measured by CD4+ count) despite failing to achieve viral suppression, or, vice versa, patients who maintain or reduce CD4+ cell count despite achieving viral suppression. Indeed, it is well known that higher CD8 activation is associated with fewer treatment-mediated CD4 gain. Each 10% increase in activated CD8+HLADR+CD38+ mean 90 fewer CD4 cell gained (Hunt PW et al J Infect Dis. 2003. 187:1534-43). The failure of recover CD4 T cells may rely on a incomplete viral suppression than could be responsible for increased immune activation and lymphocyte death. Recently, it has been pointed out that intensification strategies may be useful in reducing activation and improving CD4 T cell recovery (Kolber MA, et al, Clin Immunol. 2007 [Epub ahead of print]).

ELIGIBILITY:
Inclusion Criteria:

1. Patient having a diagnosis of HIV infection, on continuously HAART for at least 2 years, including:

   * 2 NRTI/NtRTIs (except ddI+TDF), plus
   * 1 PI/ritonavir (lopinavir/ritonavir, atazanavir/ritonavir, fosamprenavir/ritonavir, tipranavir/ritonavir, darunavir/ritonavir) or 1 NNRTI (nevirapine or efavirenz)
2. Undetectable plasma HIV-1 RNA (VL < 50 copies/mL) during the last 2 years prior to screening (with at least 4 determinations of viral load during this time period).
3. Good treatment adherence.
4. No presence of other factors which could contribute to CD4+ declines, such as treatment with chemotherapy, treatment with interferon/ribavirin, a ddI+TDF-containing regimen, etc, at least 12 months prior to screening.
5. Patient classified as "discordant" who showed high level of CD8+HLADR+CD38+ and cell death values at the screening (see reference values in the definition section in page 9: 4.2. AIMS).
6. Voluntary written informed consent.

Exclusion Criteria:

1. Pregnancy or fertile women willing to be pregnant.
2. Acute infections or uncontrolled chronic infection in the 2 months previous to the inclusion.
3. Hepatic toxicity (AST, ALT levels grade +/= 3).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
CD4 cell count | From Basal to 48 week (last visit) every 3 months

SECONDARY OUTCOMES:
Epidemiologic variables: Age, sex, time of HIV diagnosis/duration of HIV infection, duration of antiretroviral treatment with HAART, duration of treatment with a PI, HIV infection status/CDC disease stage. Epidemiologic, virologic, and immunologic data | Baseline
Virologic and immunologic variables: Time/duration of viral suppression, nadir CD4+ count, change in CD4+ count (absolute and percentage) since initiation of antiretroviral therapy, since initiation of HAART, and since achieving and undetectable viral | From Basal to 48 week (last visit) every 3 months
Apoptotic variables: Cell death in CD4 and CD8 cells, defined as the percentage of cells which present a weak DIOC measurement (DIOC low) after 1 or 4 days of culture. | From Basal to 48 week (last visit) every 3 months
The toxicity parameters will be evaluated: Hematology: Hematocrit, red blood cell count, hemoglobin, MCV, lymphocyte, platelet count, quick Index. • Biochemistry: glucose, total cholesterol, HDL and LDL cholesterol, triglycerides, urea, creatinine, A | From Basal to 48 week (last visit) every 3 months
Clinical adverse effects and clinical events | From Basal to 48 week (last visit) every 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- H.U. Germans Trias i Pujol, Badalona, Barcelona, Spain